CLINICAL TRIAL: NCT02792764
Title: A Prospective, Multi-centered Study to Assess the Complication Rates of Oncology Patients Accessed With Peripheral Intravenous Lines Versus Implantable Ports for Chemotherapy Administration
Brief Title: Post-Marketing Study to Assess Complication Rates of Oncology Patients With Ports and Peripheral IVs
Acronym: VEINSFORLIFE
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: BPV-13-003
Record Dates: First submitted 2014-04-15; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-02

CONDITIONS: PORTs/Peripheral IVs Complication Rates
Keywords: port; peripheral intravenous lines; oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Port: Subjects receiving chemotherapy through a port
- Peripheral Intravenous (PIV) Lines: Subjects receiving chemotherapy through a peripheral IV

SUMMARY:
This study is to collect current information on complications rates of subjects undergoing chemotherapy administration through Ports and peripheral IVs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 21 years
* Subject is currently undergoing or has had infusional cancer therapy (solid tumor or hematologic) through a Bard PORT with a distally-valved catheter/open-ended catheter or infusion through a PIV
* Subject had a chemotherapy regimen consisting of a vesicant and/or irritant
* Subject has signed an Informed Consent Form (ICF) or has had an ICF signed by the subject's legally authorized representative

Exclusion Criteria:

* Subject has/had an implanted non Bard PORT

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who are currently undergoing or has had infusional cancer therapy (solid tumor or hematologic) through a Bard PORT with a distally-valved catheter/open-ended catheter or infusion through a Peripheral IV
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The rate of adverse events in subjects undergoing chemotherapy administration through PORTs and PIVs. | Through end of chemotherapy, up to 3 years
  Subjects medical records will be retrospectively reviewed from present day back to January 1, 2008 to assess for complications

SECONDARY OUTCOMES:
The average number of accesses during course of treatment (i.e. - chemotherapy administration, CTs, blood draws, TPN, etc.) | Through end of chemotherapy, up to 3 years
  Subjects medical records will be retrospectively reviewed from present day back to January 1, 2008 to assess for complications
The rate of Vascular Access Device conversion from Peripheral IV to PORT | Through end of chemotherapy, up to 3 years
  Subjects medical records will be retrospectively reviewed from present day back to January 1, 2008 to assess for complications
The average time of vascular access device conversion from Peripheral IV to PORT | Through end of chemotherapy, up to 3 years
  Subjects medical records will be retrospectively reviewed from present day back to January 1, 2008 to assess for complications

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Quincy Medical Group, Quincy, Illinois
  - Willis Knighton Cancer Center, Shreveport, Louisiana

IPD SHARING:
Plan to Share IPD: No